CLINICAL TRIAL: NCT05993793
Title: Use of Fototherapy in the Treatment of Fissura in Ano
Brief Title: Use of Fototherapy in the Treatment of Fissure in Ano
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 53623621.0.0000.5544
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Fissure in Ano
Keywords: fissure; ano; phototherapy
MeSH Terms: conditions — Fissure in Ano

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fototherapy (Experimental)
  Interventions: Device: Fototherapy

INTERVENTIONS:
Device: Fototherapy — The Antares brand Laser device was used for 3 sessions with an interval of 24 hours. The Visual Analogue Scale (VAS) was used before starting treatment, after the first and second sessions, and 1 week after the third session. In addition, at the end of the treatment, the closure, or not, of the lesion was verified, and the questionnaires performed prior to phototherapy were reapplied. The VAS assesses the patient's level of pain, which can be divided into mild pain (1-2), moderate pain (3-7), and severe pain (8-10). The Bristol Scale is based on the identification of the patient's consistency of stools, while types 1-2 correspond to constipation, 3-4 indicate normal intestinal rhythm, 5 indicate lack of fiber, and 6-7 correspond to diarrhea

SUMMARY:
The eligible population consisted of individuals with anal fissure awaiting surgical intervention. Individuals aged 18 years or older were included, diagnosed with anal fissure and who voluntarily agreed to participate in the research. Those who had some pelvic inflammation and who had already undergone a surgical procedure and had recurrence were excluded from the studyThe selected individuals underwent a standardized anamnesis of the service, answered questionnaires on symptoms of intestinal constipation (Rome IV Criteria and the Bristol Scale), underwent a physical evaluation by a trained professional, and then began the application of the research protocol. The Antares brand Laser device was used for 3 sessions with an interval of 24 hours. The Visual Analogue Scale (VAS) was used before starting treatment, after the first and second sessions, and 1 week after the third session. In addition, at the end of the treatment, the closure, or not, of the lesion was verified, and the questionnaires performed prior to phototherapy were reapplied. The VAS assesses the patient's level of pain, which can be divided into mild pain (1-2), moderate pain (3-7), and severe pain (8-10). The Bristol Scale is based on the identification of the patient's consistency of stools, while types 1-2 correspond to constipation, 3-4 indicate normal intestinal rhythm, 5 indicate lack of fiber, and 6-7 correspond to diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* individuals with the diagnosis of anal fissure that accepted to participate as volunteers in the clinical trial

Exclusion Criteria:

* individuals with pelvic inflammation
* individuals who have been through surgical procedures
* individuals who have relapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Complete closure of the fissure | 15 days
  It is estimated that the fototherapy will close completely the fissure in patients with fissure in ano.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Patrícia Lordelo, Salvador, Estado de Bahia, Brazil